CLINICAL TRIAL: NCT04870398
Title: Treatment Outcome of Partial Pulpotomy by Using Two Different Bioactive Materials in Mature Permanent Teeth With Signs and Symptoms of Irreversible Pulpitis. A CONSORT Randomized Clinical Trial
Brief Title: Partial Pulpotomy in Mature Permanent Teeth With Signs and Symptoms of Irreversible Pulpits
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Giorgos Tzanetakis, Assistant Professor, National and Kapodistrian University of Athens
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 459/01.03.2021
Record Dates: First submitted 2021-04-24; First posted 2021-05-03 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Irreversible Pulpitis

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MTA partial pulpotomy (Active Comparator): Profound local anesthesia of the tooth and the surrounding tissues will be achieved The tooth will be isolated with a rubber dam and initial caries removal will be performed by using a sterile high speed diamond bur. The deeper layers of caries will be removed by using a series of different diameters sterile low speed burs. After complete caries removal and pulp tissue exposure, first cut of pulp tissue will be performed using a new sterile high speed diamond bur. After the inspection of the surgical field for residual caries and the irrigation of the cavity with physiologic saline solution, a sterile cotton pellet will be gently placed over the pulp tissue for 3 minutes. Once hemostasis is achieved, a blood-filled homogenous tissue without dark or yellowish areas will be considered essential for the placement of MTA. After the placement of MTA, a resin modified glass-ionomer cement will be placed over the capping material and the cavity will be sealed with resin-bonded composite
  Interventions: Procedure: Vital Pulp therapy-Partial pulpotomy
- Total Fill partial pulpotomy (Active Comparator): The tooth will be isolated with a rubber dam and initial caries removal will be performed by using a sterile high speed diamond bur. The deeper layers of caries will be removed by using a series of different diameters sterile low speed burs. After complete caries removal and pulp tissue exposure, first cut of pulp tissue will be performed using a new sterile high speed diamond bur. After the inspection of the surgical field for residual caries and the irrigation of the cavity with physiologic saline solution, a sterile cotton pellet will be gently placed over the pulp tissue for 3 minutes. Once hemostasis is achieved, a blood-filled homogenous tissue without dark or yellowish areas will be considered essential for the placement of Total Fill BC. After the placement of the material, a resin modified glass-ionomer cement will be placed over the capping material and the cavity will be sealed with resin-bonded composite
  Interventions: Procedure: Vital Pulp therapy-Partial pulpotomy

INTERVENTIONS:
Procedure: Vital Pulp therapy-Partial pulpotomy — Removal of inflamed pulp tissue, hemostasis and placement of pulpotomy material

SUMMARY:
The main purpose of the present study is to assess the outcome of partial pulpotomy by using two different bioactive materials, namely MTA [MTA Angelus (Angelus, Londrina, Brazil) and Total Fill BC putty (FKG, La Chaux-de-Fonds, Switzerland) bioceramic material in mature teeth with deep caries and clinical symptoms indicative of irreversible pulpitis. A secondary aim is to evaluate whether age, tooth type and coronal restoration play a significant role on the outcome of partial pulpotomy in the evaluated cases.

DETAILED DESCRIPTION:
Study design This is a randomized controlled clinical superiority trial, parallel designed which will be conducted in compliance with the CONSORT and PRIRATE 2020 guidelines for reporting randomized trials in Endodontology recently published by the ESE (Nagendrababu et al. 2020a, b). During the study, two different bioactive materials will be tested upon their placement on exposed pulps of mature teeth with preoperative signs and symptoms indicating the presence of irreversible pulpitis. Patients referred to the Postgraduate Clinic of Endodontology of Dental School of National and Kapodistrian University of Athens, will participate in the study.

Sample size calculation For sample size calculation, the Stata version 15.1 software (Stata Corp, College Station, Texas, USA) has already been used. Based on the results of a previous study by Taha & Khazali (2017) and expecting a 85% success rate for tested materials with 80% power of analysis and determining the level of statistical significance at 5%, the number of patients in each group was determined to be 65 (n = 65).

Randomization/Allocation concealment/Bliniding The randomization of the patients in the study has been taken place by using the web-based software of www.randomizer.org. This software gives automatically numbers to patients allocating them randomly in the study groups. Patients will be blinded to the type of the material used in their tooth. The operator could not be blinded during the study. An experienced endodontist (more than 15 years of clinical experience) will assess the follow-up radiographs and will be blinded to the capping material used in each case.

Data collection Demographic data such as age and sex and data regarding the tooth type and location will be collected.

Preoperative clinical and radiographic examination At the first appointment, the medical and dental history including the chief complaint will be recorded and then clinical and radiographic examination will take place. Accurate history of pain will take place to assess the severity of pain including the spontaneity or the lingering of pain after temperature stimulation and the sleep disturbance. The patients that meet the inclusion criteria will be informed in details about the aims of the study and those who will give permission will sign an informed consent and will be added to the study with a recognition number.

Clinical examination will consist of:

* Visual inspection of the caries lesion under operating microscope.
* Restorability of the tooth.
* Percussion and palpation tests.
* Cold and electric pulp sensibility tests.
* Periodontal examination (pocket depth, attachment loss and mobility). A clinical diagnosis indicating the establishment of irreversible pulpitis will be set in all cases based on the history of severe spontaneous or lingering pain reproducible during clinical examination.

Radiographic examination Preoperative periapical radiographs will be taken using the parallel cone technique using the Rinn set. (Rinn, Dentsply, Elgin, IL).

Clinical Intervention All the procedures will be carried out by the same experienced operator (GT, more than 15 years of clinical experience in his practice limited to Endodontics) and under operating microscope by using high magnification. High quality photographs will be taken throughout the procedures. Profound local anesthesia of the tooth and the surrounding tissues will be achieved by using lidocaine with 1/80000 epinephrine (Lignospan Special, Septodont, France). The tooth will be isolated with a rubber dam and initial caries removal will be performed by using a sterile high speed diamond bur. The deeper layers of caries will be removed by using a series of different diameters sterile low speed burs. After complete caries removal and pulp tissue exposure, first cut of pulp tissue will be performed using a new sterile high speed diamond bur. After the inspection of the surgical field for residual caries and the irrigation of the cavity with physiologic saline solution, a sterile cotton pellet will be gently placed over the pulp tissue for 3 minutes. If bleeding continues after the removal of cotton pellet, NaOCl 2.5% will be used for irrigation of the pulp tissue and a new sterile cotton pellet will be placed over the pulp for another 2 minutes. In case where bleeding continues after the removal of the new cotton pellet, a second cut of the pulp tissue will be performed to reach a tissue free of inflammation. Then, a new sterile cotton pellet will be placed over the amputated pulp for 5 minutes. If bleeding continues, the case will be excluded from the study and full pulpotomy or root canal treatment will be considered. Once hemostasis is achieved, a blood-filled homogenous tissue without dark or yellowish areas will be considered essential for the placement of pulp capping material. All the materials tested will be prepared according to the manufacturers' instructions. After the placement of the materials, a resin modified glass-ionomer cement (Ultrablend Plus, Ultradent Products Inc.) will be placed over the capping material and the cavity will be sealed with resin-bonded composite (Estelite Quick, Tokuyama Dental, Tokyo, Japan). A telephone call will be scheduled with the patient after one, two, three and four days in order to get information about the clinical condition of the tooth, the pain relief and the anti-inflammatory drugs needed postoperatively. In case of severe pain persisting one week after the intervention, the patient will be scheduled for root canal treatment and the case will be recorded as clinical failure.

Recall protocol Follow-up clinical and radiographic examinations are scheduled at 3, 6, 12, 24, 36 and 48 month intervals. A dental history will be obtained, including possible pain experience or pain and discomfort during mastication as well as the functionality of the tooth. The teeth will also be clinically examined for signs and symptoms such as pain or discomfort during percussion, swelling or sinus tract, presence of periodontal pocket and absence of positive response to cold testing. Radiographic examination will include the assessment of periapical status, the formation of dentin bridge and the presence of internal resorption or root canal obliteration. Finally, the quality of coronal restoration will be assessed clinically and radiographically.

Statistical analysis Descriptive statistics with cross tabulations will be performed. Baseline characteristics of the sample will be tabulated and frequency distributions will be presented for all covariates (sex, age, type of tooth, dentin bridge formation, type of coronal restoration), across type of pulp capping material. Chi-squared and Fisher's exact tests will be applied as appropriate. Kaplan-Meier survival curves for pulp capping materials, type of tooth, age band and sex will be also drawn. Log-rank tests for equality of survivor functions will be applied. A univariable and multivariable random effects Cox regression model, using the date of entry to the study as the time-scale, will be built based on pre-defined covariates, such as pulp capping material, tooth type, sex, age, dentin bridge formation and type of coronal restoration. All predictors will be retained in the final multivariable model. The proportional hazards assumptions will be checked through Nelson Aalen plot for log cumulative hazard by type of pulp capping material. A two-sided p-value of 0.05 will be used to determine statistical significance for all analyses, along with 95% CIs. All analyses will be performed using Stata v.14.1.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 10 years old.
* Written consent after their update regarding the study and its aims.
* Noncontributory medical history.
* Extremely deep caries extending to the pulp chamber.
* Positive response to cold sensibility testing.
* Presence of spontaneous pain or provoked lingering pain to cold stimuli.
* No clinical signs of pulp necrosis such as swelling or presence of a sinus tract.
* Restorable and periodontally sound teeth.

Exclusion Criteria:

* Immature teeth.
* Cariously involved teeth with no response to pulp sensibility tests.
* No signs and symptoms of irreversible pulpitis.
* Bleeding not controlled in 10 minutes after partial pulpotomy.
* Teeth with no evidence of bleeding after communication with the pulp chamber (necrosis of the coronal pulp tissue)
* Teeth with the pulp chamber exposed to the oral environment.
* Detection of periodontal pocket with depth greater than 4mm.
* Teeth suspected for crack or incomplete crown fracture possibly responsible for pulp pathology.
* Medically compromised patients.

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2017-01-05 (Actual); Primary Completion 2021-04-23 (Actual); Study Completion 2021-04-23 (Actual)

PRIMARY OUTCOMES:
Number of successful cases with vital and healthy pulp during the follow-up period | 1-4 years
  The primary outcome will be defined clinically in the absence of pathologic signs and symptoms such as spontaneous or lingering pain, tenderness to percussion and swelling as well as the response to cold sensibility test. Radiographically, the assessment of periapical tissues will take place. If the periapical tissues were normal preoperatively, they should continue to be normal. If a periapical radiolucency was present preoperatively, then a complete healing of periapical tissues should be accomplished. Under the above conditions, the case will be considered successful. If a case presents severe spontaneous or lingering pain, tenderness or pain to percussion, swelling or sinus tract with persistence of periapical lesion or emergence of a new one, will be considered as failure.

SECONDARY OUTCOMES:
Assessment of pain after pulpotomy procedure using the Heft-Parker visual analog scale | One week after the intervention
  The secondary outcome of pain after intervention will be assessed through the recall examination of each patient one week postoperatively. Each patient will be asked if he/she experienced or not pain postoperatively and in case of postoperative pain, he/she will be asked about the duration and the characteristics of the pain and if anti-inflammatory drugs were needed for pain control. Intensity of pain will be assessed by using the Heft-Parker visual analog scale

CONTACTS AND LOCATIONS:
Overall Officials: Giorgos N Tzanetakis, Principal Investigator — Department of Endodontics, School of Dentistry, National and Kapodistrian University of Athens

IPD SHARING:
Plan to Share IPD: Yes
Study protocol and Statistical analysis plan
Supporting Information: Study Protocol, SAP
Time Frame: Ever
Access Criteria: Partial pulpotomy